CLINICAL TRIAL: NCT05751369
Title: The Tobacco, E-Cigarette, and Cannabis Waste Randomized Controlled Trial
Brief Title: Addressing Tobacco, E-Cigarette, and Cannabis Waste
Acronym: TECW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Marcos (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1896205; T321R4972 (Other Grant/Funding Number: California Tobacco Related Disease Research Program)
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Educational Status; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education Only (Active Comparator): Treatment as usual with brief videos and weblink
  Interventions: Behavioral: Education plus Support
- TECW+ (Experimental): Education plus motivational enhancement
  Interventions: Behavioral: Education plus Support

INTERVENTIONS:
Behavioral: Education plus Support — Brief behavioral support for using TECW Tracker
  Other Names: Motivational Enhancement

SUMMARY:
This study tests of effect of brief education and support about tobacco, e-cigarette, and cannabis waste (TECW) on knowledge, beliefs, behavior, and TECW on two college campuses.

ELIGIBILITY:
Inclusion Criteria:

* student at University of California, Davis or California State University San Marcs
* between the ages of 18 and 25
* taking at least one class on the main campus
* at least six months until graduation
* have a smart phone with location services enabled for apps
* regular access to a device with sufficient WiFi
* private space for three remote visits on over the next six weeks and one visit in six months
* willing to have camera on during remote visits

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
Knowledge about TECW | 6 weeks
  Percent correct on 12-item knowledge test based on Protect our Planet: The Earth is Not Disposable (California Youth Advocacy Network) and Environmental Impact of Cigarette Butts (Tobacco Free CA) videos. Higher scores reflect more accurate knowledge about TECW

SECONDARY OUTCOMES:
Perceived harmfulness of TECW | 6 weeks
  Questions adapted from Epperson et al. (2021) and Hoek et al. (2020); score ranges from 1-5, higher scores reflect greater perceived harm
Belief that TEC manufacturers should be accountable for waste mitigation | 6 weeks
  Questions adapted from Hoek et al. (2020); score ranges from 1-4, higher scores reflect stronger regulatory belief
Use of TECW Tracker | 6 weeks
  Number of reports received in ArcGIS-based TECW Tracker program
Readiness to engage in regulatory behavior | 6 weeks
  Questions adapted from Pulvers (2022); scores range from 1-5; higher scores reflect greater regulatory readiness

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - California State University San Marcos, San Marcos, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pulvers K, Nordskog AB, Shearer H, Smith C, Stewart SL, Novotny TE, Tong EK. Modifying Tobacco and Cannabis Waste Perceptions and Behavior Among Young Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 4;14:e79525. doi: 10.2196/79525. PMID 41343823